CLINICAL TRIAL: NCT04410471
Title: Development and Persistence of Humoral Immunity Against SARS-CoV-2 in Liver Transplanted Patients in Comparison With Immunocompetent Patients
Brief Title: Humoral Immunity Against SARS-CoV-2 in Liver Transplanted Patients After COVID-19 in Comparison With Immunocompetent Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Magdalena Salcedo (Other)
Responsible Party: Sponsor-Investigator, Magdalena Salcedo, Attending Physician, Hepatology, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: Sero-Covid19_TH
Record Dates: First submitted 2020-05-29; First posted 2020-06-01 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Liver Transplant Infection; Covid19; Mortality; Immune Response
Keywords: Humoral Immunity; Reinfection; IgG and IgM against SARS-CoV-2; Immunosuppression
MeSH Terms: conditions — COVID-19; Reinfection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Liver transplant patient after having Covid19: Adult Liver transplant patient who had survived to Covid19 in the first wave of the disease in Spain (disease until june 30th), in all the liver Transplant Units in Spain (24).
  Interventions: Diagnostic Test: CLIA of IgG and IgM against SARS-Cov-2
- No immunosuppressed patient with previous Covid19: Not immunosuppressed patient who had survived to Covid19 in the first wave of the disease. These patient have been diagnosed and treated in the Hospital Gregorio Marañón (Madrid), before 30th June
  Interventions: Diagnostic Test: CLIA of IgG and IgM against SARS-Cov-2

INTERVENTIONS:
Diagnostic Test: CLIA of IgG and IgM against SARS-Cov-2 — Report of clinical data
  Other Names: Nasopharyngeal PCR test of SARS-Cov-2

SUMMARY:
This is a prospective study analyzing the development of humoral immune response against SARS-Cov-2 in patients with previous Covid19: the aim is to compare the incidence, titration and evolution of IgG an IgM in a prospective cohort of liver transplant patients surviving to the first wave of Covid19, in comparison to not inmmunossupressed patients.

DETAILED DESCRIPTION:
The liver transplant (HT) recipient population is more susceptible to infections than the general population. Few data are available regarding the incidence and clinical course of SARS-CoV-2 infection in this population, initially considered to be "high risk" regarding a possible higher incidence and severity of infection in these patients.

A prospective cohort of liver transplant recipient patients diagnosed with SARS-CoV-2 infection (Clinical Trials.gov Protocol Record HCB / 2020/0384) has been developed from SETH (Spanish Society for Liver Transplantation). This study aims to analyze the incidence and establish the clinical evolution of the infection in these patients. Initial data from the cohort, which includes 111 incidental cases diagnosed as of April 7, show a higher standardized incidence than the general population, but not higher mortality (data being published).

The chronic immunosuppression in t solid organ transplant patients could play a double role with respect to SARS-Cov-2 infection: on the one hand, it may condition a greater susceptibility and initial aggressiveness, in relation to itself viral effect, and in the other hand, it could protect by reducing the immune response that triggers the pulmonary and systemic inflammatory process.

After the initial Covid-19 outbreak, both in the general population and in immunosuppressed patients, the rate of specific IgM and IgG seroconversion against this coronavirus, and its protective capacity against reactivations or reinfections, are unknown. Therefore, it is a challenge for health organizations to identify the immune response in the population and to characterize its degree of protection, to adopt early measures to lessen the consequences of possible epidemic waves in the coming months.

Continuing with the prospective study of the cohort of liver transplant patients diagnosed with Covid-19 (SETH-Covid-19), already defined and composed of 91 living patients, the humoral immune response and its evolution in the first 12 months after initial infection. The cohort will incorporate the new incidental cases; A comparative study will be carried out with a contemporary cohort of non-immunosuppressed patients, controlled for age, gender and severity of the initial disease.

ELIGIBILITY:
Inclusion Criteria:

Patients recovered of covid 19 Informed Consent

Exclusion Criteria:

Chemotherapy on going Concomitant Autoimmune diseases

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Liver transplant and control patients (propensity score including age, sex, and severity of previous covid19 episode)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of IgG against SARS-CoV-2 | one year
  Proportion, Rate

SECONDARY OUTCOMES:
titration and evolution of humoral response (IgG) along first 12 months after having Covid-19 | 12 months
  Titer
Reinfection of Covid-19 | one year
  Categoric Yes/Not

OTHER OUTCOMES:
Mortality | 12 months after Covid-19
  Rate

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Salcedo, MD PhD, Principal Investigator — Liver Transplantation Unit
Locations (2):
- Spain (2):
  - Victor Fernandez Alonso, Madrid
  - Victor Fernández Alonso, Madrid

IPD SHARING:
Plan to Share IPD: Undecided
Multicenter study